CLINICAL TRIAL: NCT06783205
Title: Does Restriction of the Dominant Hand Due to Injury Improve Non-Dominant Hand Function?
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sedanur Güngör, Principal Investigator, Gazi University
Other Study IDs: 2024-390
Record Dates: First submitted 2025-01-13; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Dexterity; Tendon Injuries; Fractures; Nerve Injury
MeSH Terms: conditions — Tendon Injuries; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with orthosis/cast: Patients referred to the Hand Rehabilitation Unit of Gazi University, Faculty of Health Sciences, for physiotherapy and rehabilitation due to hand-related pathologies, and who meet the inclusion and exclusion criteria, will be informed about the study. No treatment other than routine care will be administered. Only two evaluations will be conducted: one at the first session and the other at the end of the 6th week.
  Interventions: Other: Restriction of the Dominant Hand Due to Splint Use

INTERVENTIONS:
Other: Restriction of the Dominant Hand Due to Splint Use — This study aimed to assess whether the non-dominant hand function changes in patients using splints or casts on their dominant hand during the tissue healing period.

SUMMARY:
Hand injuries result in the restriction of use of the injured hand within a splint or a plaster during the first 6 weeks which is critical for tissue healing. When the dominant hand is injured, patients experience more difficulty in daily life due to this restriction. Patients injured on their dominant hand mostly express that they are forced to use their non-dominant hand in their activities and as a result, the function of the non-dominant hand improves. However, the non-dominant hand function has not been analyzed in patients with restricted use of the dominant hand during the tissue healing period.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who need to use a splint for 6 weeks due to any pathology in their dominant hand
* Ages between 18-65
* Individuals who are within the first 10 days after the operation

Exclusion Criteria:

* Individuals with an isolated thumb injury
* Those who require bilateral use of the splint/have bilateral pathology
* Those who have a condition that prevents the use of the non-dominant hand
* Those who can use both hands equally/do not have a dominant side (ambidextrous/two-handed)
* Those who have a cooperative status that will not comply with the treatment program
* Data from individuals who do not use the splint as described during the 6-week follow-up period will not be included in the analysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Hand Rehabilitation Unit of Gazi University, Faculty of Health Sciences, for physiotherapy and rehabilitation due to hand-related pathologies, and who meet the inclusion and exclusion criteria will be included.
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2024-04-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
hand function | 6 weeks
  Hand function will be assessed using the Jebsen Taylor Hand Function Test (JTHFT), a valid tool for evaluating impairment and disability. The test includes tasks involving common grip types in daily life, aiming to measure the speed of task performance. Standardized materials, easily available in clinics, are used. The test has seven tasks: writing a 24-letter text, turning cards, collecting small objects, eating, stacking checkers, collecting light wide objects, and collecting heavy wide objects. A 1-minute rest is given between tasks, and completion time is recorded in seconds. Before evaluation, examples will be provided, and individuals will perform a trial run of each task. In our study, only the unaffected, non-dominant hand will be assessed, starting with a single real assessment after the trial.

SECONDARY OUTCOMES:
disability level | 6 weeks
  Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire will be measured. This questionnaire is used to assess upper extremity disorders and includes 30 items covering pain, stiffness, weakness, daily activities, and functionality. Patients consider their condition over the past week, with total scores ranging from 0 to 100. Higher scores indicate worse functional status.
Grip and pinch strengths | 6 weeks
  Gross grip strength will be measured with a hydraulic hand dynamometer (Jamar®) and fine grip strength with a pinchmeter. Participants will sit in a chair with back support, following the standard position: arm at the side, elbow at 90° flexion, and wrist neutral. Fine grip strength will be assessed in double (bipod) pinch, triple (tripod) pinch, and lateral grip positions. The forearm will be fully pronated for double and triple pinches, and midpronated for gross grip and lateral grips. Only the healthy non-dominant hand will be assessed. Measurements will be repeated three times, and participants will squeeze as hard as possible. The average of the three trials will be recorded in kilograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Health Science Faculty Physiotherapy and Rehabilitation Department, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided